CLINICAL TRIAL: NCT02112942
Title: A Phase I Study Assessing Single and Multiple Doses of IDX21459 in Healthy and HCV-Infected Subjects
Brief Title: Study Assessing Single and Multiple Doses of IDX21459 in Healthy and HCV-Infected Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Early termination of IDX21459 was due to integration of Merck's HCV antiviral pipeline has resulted in revisions of the clinical development plan.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7822-001; IDX-04C-001
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C virus; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Healthy subjects, sequential dose escalation, IDX21459 capsules or Matching Placebo capsules, once daily, up to 7 days
  Interventions: Drug: IDX21459; Drug: Matching Placebo
- Group B (Experimental): HCV subjects genotype 1, IDX21459 capsules, once for 1 day
  Interventions: Drug: IDX21459
- Group C (Experimental): HCV subjects genotype 1, IDX21459 capsules or Matching Placebo capsules, once daily, for 7 days
  Interventions: Drug: IDX21459; Drug: Matching Placebo

INTERVENTIONS:
Drug: IDX21459
Drug: Matching Placebo
  Arms: Group A; Group C

SUMMARY:
A multi-part study to evaluate the safety and PK of single ascending doses of IDX21549 in healthy and HCV-infected subjects. The effect of food on the PK of IDX21549 will also be evaluated. Antiviral activity will also be assessed in HCV-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Subjects are in good general health.
* Subjects have provided written informed consent form.
* All subjects of childbearing potential must have agreed to use a double method of birth control (one of which must be a barrier) from Screening through at least 90 days after the last dose of the study drug. HCV Subjects
* Documented clinical history compatible with chronic hepatitis C without cirrhosis.
* Treatment-naïve
* HCV Genotype 1

Exclusion Criteria:

All subjects

* Pregnant or breastfeeding
* Co-infected with hepatitis B virus (HBV) and/or human immunodeficiency virus (HIV).
* Decompensated liver disease
* Other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessment | up to 35 days
  Proportion of subjects experiencing adverse events.

SECONDARY OUTCOMES:
Pharmacokinetic | Up to 120 hours post dose
  Plasma and urine concentrations of IDX21459 and its metabolite/s.